CLINICAL TRIAL: NCT03763383
Title: Lateral Arm Flap: Usage as Pedicle and Free Flap :A Case Series
Brief Title: Lateral Arm Flap Usage as Pedicle and Free Flap
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Sami Ullah, Sami Ullah (principal investigator), Aga Khan University
Other Study IDs: lateral arm
Record Dates: First submitted 2018-11-16; First posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Flap Necrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Free lateral arm flap: included patients who had free lateral Arm flap
  Interventions: Procedure: Lateral Arm Flap
- pedicled lateral arm flap: included patients who had pedicled lateral arm flap
  Interventions: Procedure: Lateral Arm Flap

INTERVENTIONS:
Procedure: Lateral Arm Flap — Its a kind of flap that is harvested from the lateral aspect of the arm to cover defects in different parts of the body

SUMMARY:
Abstract

Introduction For local reconstruction on upper extremity or as a distant micro vascular flap Lateral arm free flap is an excellent source of tissue with the advantages including short operation time, thin pliable tissue, non-dominant vessel and minimal donor site morbidity, it fulfills the goal of an optimal reconstruction of form, function, and aesthetics .Here the investigator share his experience of lateral arm fasciocutaneous flap, investigator found it effective in covering defects secondary to trauma, malignancy and burns.

Methods A retrospective data analysis was done to analyze our usage of lateral arm flap. This included patient's age, sex, primary problem, area involved, size of the flap and outcome of the flap 3 weeks post operatively. For free flaps this also included the recipient artery used for anastomosis and the number of veins anastomosed.

Results There were 21 flaps done over a period of five years. This included 11 free flaps and 10 pedicle flaps. Average size of free flap was 12x5 cm and that of pedicle flap was 8x5 cm. In the free flap group, there was failure in 2 flaps both of which were due to arterial anastomoses in zone of injury. In the pedicle flap group however, there were no failures.

Conclusion Lateral arm flap is a reliable flap with consistent anatomy that can be used for coverage in different parts of the body.

DETAILED DESCRIPTION:
1. Introduction One aspect of reconstructive surgery is to replace any lost tissue with similar tissue. With advent of microsurgery it is now possible to achieve better aesthetic results with reduced donor site morbidity.

   For soft tissue replacement, Radial Forearm Flap had been the procedure of choice since its description in Chinese literature. Problems associated with Radial forearm flap included donor site morbidity and loss of major artery of forearm. This was replaced by anterolateral thigh flap that was described by Song et al in 1984 1 and popularized by Fu Chan Wei. 2 However, its drawback comprises of it being a bulky flap.

   Lateral arm free flap was first described by Katsaros et al 3 is a versatile free flap, which can be used in many reconstructions and is now commonly used in upper extremity reconstruction both as a reverse pedicle and as a free flap. It is well suited to cover defects where a thin flap is required especially dorsum of the hand.3, 4, 5 Having advantage of being thinner than the anterolateral thigh flap it also does not sacrifice a major artery and has acceptable donor site morbidity. However, its drawback includes a shorter pedicle and smaller skin paddle. 6

   Here investigator share his experience of using the lateral arm flap both as a free flap and as a pedicle flap.
2. Materials and Methods A retrospective review of 21 patients who underwent lateral arm flap reconstruction for various defects in the body from January 2012 to December 2016 was carried out. Patients were grouped into two main categories and were followed for 3 weeks post operatively .Group 1 included patients who had Free Lateral Arm Flap (FLAF), Group 2 included those who had reconstruction using Pedicle Lateral Arm Flap (PLAF). Data was collected using a standard Performa containing details about patient's age, sex, etiology of defect, area involved, size of flap and outcome (survival/failure) of the flap. For free flaps, this also included the recipient vessels used for anastomosis and the number of veins anastomosed. The work has been reported in line with the PROCESS criteria.7

4. Operative Procedure: Operative procedure was the same as described in literature. 7 The vascular supply of the lateral arm flap is the posterior radial collateral artery (PRCA) which is the branch of the radial collateral artery. The PRCA runs in the lateral intermuscular septum of the arm. A line drawn from the deltoid insertion to the lateral epicondyle denotes the lateral intermuscular septum. (Fig 1 a) Anteriorly, the intermuscular septum is bounded by brachialis and brachioradialis and posteriorly by the triceps. If ELAF extended lateral arm flap is required then a line is drawn from the lateral epicondyle to the radial styloid.

4.1. Reverse flap: The vascular supply of this flap is based on the epicondylar and olecranon plexi which are supplied by the interosseous recurrent artery IRA and the radial recurrent artery RRA.

While harvesting the flap, posterior incision is made first. The triceps muscle is identified and intermuscular septum is reached. (Fig 1 b) Here perforators from the PRCA are identified. For ELAF it is necessary to identify a perforator 4 cm above the lateral epicondyle. Once the perforators are identified the main vessel is identified in the septum and elevated from above the periosteum of the humerus. If a reverse flap is required then the distal anastomosis is kept intact and the vessel is divided proximally.

If a free flap is required the vessel is traced proximally to the main vessel. Here while ligating the anterior radial collateral artery ARCA radial nerve needs to be protected. Once adequate vessel length has been achieved the anterior incision is given. Once flap is elevated it is left to bleed for at least 15 minutes before division.

Figure 1:

a. Marking of flap b Elevated flap. Triceps muscle can be seen posteriorly and Radial nerve coursing above it.

5. Case 1

A 32 year old male presented with trauma to right hand dorsum which was entrapped in a generator belt. (Fig 2) He had loss of extensor tendons of second and third digit secondary to fractured second metacarpal. Initially he had two debridements in which the bone was fixed with a k wire. He then had one stage reconstruction of the defect. First, plantaris tendon graft was taken to reconstruct the extensor tendons of the second and third digits followed by lateral arm free flap measuring 11x6 cm. Arterial anastomosis was done end to side to radial artery and venous anastamoses was done to cephalic vein and venae comitantes. He did well postoperatively and recovered all his functions.

Figure 2:

a Wound at presentation b Flap coverage

6. CASE 2 A 33 years old female presented with a history of burns in 1994. (Fig 3) She presented to us 19 years later with post burn contractures involving the neck, chest and bilateral axilla. Neck contracture involved upto 2/3rd of the anterior neck with a pull on the left side of the lower lip. No extension was possible however she could flex her neck. Surgical procedure involved release of neck contracture followed by reconstruction with a free extended lateral arm flap measuring 18x8cms. Artery was anastomosed end to end using superior thyroid artery and both the venae comitantes were anastomosed end to end with tributary of internal jugular vein and end to side with internal jugular vein. Contractures involving other areas were managed with ancillary procedures.

Figure 3:

1. Preop Presentation b) Intraop After Release of Contracture
2. Marking d) Follow up Two Weeks

   7. Case 3 28 year old female who had presented to us with a scar on the dorsal aspect of the forearm.(Fig 4) The patient had a lesion at the same site which was present there for about a year. On excisional biopsy the histopathology of the lesion revealed a Dermatofibrosarcoma Protuberance so she was planned for wide local excision of the scar and a free lateral flap. The defect arising upon excision of the lesion was 10x6cm which was covered with a free lateral flap of the same size. Arterial anastomosis was carried out end to end with radial artery; one vein was anastomosed end to end with venae comitantes of radial artery and the other with cephalic vein.

Figure: 4

a) Scar Pre op b) Markings for Excision

c) Flap Marking d) 1.5 years Post op

8. Discussion The free lateral arm flap provides a good option for reconstruction of simple and complex multistructural defects of small to medium size at different parts of the body. The flap has constant anatomy and relatively longer vascular pedicle besides the great variety of tissue components that are included. Change of position during surgery is usually not necessary, and the operation time can be lowered by simultaneous working of two teams. The rate of revision, complication, or flap loss is low. Secondary debulking procedures are usually not necessary on a frequent basis. A primary closure of the donor defect is worth aspiring to for an aesthetically satisfactory result.8 Since its description there have been a number of modifications in the lateral arm flap. Extended lateral arm flap (ELAF) can be harvested by designing the flap distal to the lateral epicondyle along the axis from the lateral epicondyle to radial styloid.9This modification not only increases the length of the flap but also allows for increased length of the pedicle. In this series there were two cases in which ELAF was used.

Other modifications include harvesting a cortex of the humerus, triceps muscle tendon and posterior cutaneous nerve of the forearm along with the flap.10All these modifications lead to variety of defects being reconstructed with lateral arm flap.

Another important variation of Lateral Arm Flap is Pedicle Reverse Lateral Arm Flap. Inappropriate or inadequate treatment of full-thickness wounds involving the cubital fossa inevitably results in flexion contractures and causes various degrees of restriction in the extension of the elbow joint. Once the contracture develops, restoration of full extension in the elbow joint becomes a major challenge for reconstructive surgeons. Release of contracture discloses a big skin defect that should be replaced with skin of similar nature, pliable and elastic, because of wide range of motion of the elbow joint. It is well known that there are many useful surgical techniques for resurfacing the defects around the elbow joint, including skin grafts, local fasciocutaneous flaps, local muscle flaps with or without skin, local adipofascial flaps, distant flaps and free flaps.

Local fasciocutaneous flaps have widely been used for covering the defects around the elbow joint. Pedicle reverse lateral arm flap provide stable soft tissue coverage in conjunction with a consistent axial pedicle, relative ease of dissection, and without the sacrifice of a major distal vessel, despite significant soft tissue and bony elbow trauma.13 With careful preoperative planning, this flap is a safe and reliable method of reconstruction for complex elbow injuries, though many studies described it prone to complications because of unreliable blood supply in traumatic elbow injuries. The flap was used in three patients with acute traumatic wounds on the elbow in our series without any complication.

One of the most important factor in choosing an appropriate flap for a particular defect is donor site outcome. Klinkenberg et al has mentioned that knowledge of postoperative donor-site morbidity helps in decision making in case more than any of the flaps matches the recipient-site requirements. In addition, differences concerning donor-site morbidity evaluated in their study could outweigh differences in color, texture, thickness, and hairiness of the transplanted free flap.11There have been mixed reports with respect to donor site outcome of the lateral arm flap. In a retrospective survey, Graham et al analyzed the donor site morbidity of 123 LAF and found the appearance of the scar on the lateral arm to be the major reason for dissatisfaction.12 This was especially the case when skin grafts were used to cover the donor site and when patients were females. The second major problem was reported to be the lateral epicondylar pain. These findings confirmed by other group that had also reported sensory disturbances of the lateral proximal forearm (hypoesthesia, paresthesia, and hyperesthesia), delayed wound healing, and tendon exposure to be the major complications following LAF harvest.

In contrary to the findings of Graham et al Depner et al found scar visibility to be well accepted by the patients in their study with no differences regarding gender. A possible reason for this discrepancy according to them could be related to the fact that they prefer to avoid skin grafting of the donor-site defect by limiting the flap width to 6 or 7 cm and thereby allowing primary wound closure.13 We achieved primary closure of the donor site in all patients. Two of the patient had flap width greater than 6cm however because of the larger arm circumference the donor site was closed primarily. None of the patient complained about the donor site despite the fact that one patient had donor site dehiscence.

ELIGIBILITY:
Inclusion Criteria:

1. patients who underwent free Lateral Arm Flap
2. Patients who underwent pedicled Lateral arm flap -

Exclusion Criteria:

* No specific exclusion criteria

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Flap survival/necrosis | 3 weeks
  was assessed by clinical examination noticing color and bleeding by needle prick

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Song YG, Chen GZ, Song YL. The free thigh flap: a new free flap concept based on the septocutaneous artery. Br J Plast Surg. 1984 Apr;37(2):149-59. doi: 10.1016/0007-1226(84)90002-x. PMID 6713155
- [Background] Wong CH, Wei FC. Anterolateral thigh flap. Head Neck. 2010 Apr;32(4):529-40. doi: 10.1002/hed.21204. PMID 19672962
- [Background] Katsaros J, Schusterman M, Beppu M, Banis JC Jr, Acland RD. The lateral upper arm flap: anatomy and clinical applications. Ann Plast Surg. 1984 Jun;12(6):489-500. doi: 10.1097/00000637-198406000-00001. PMID 6465806
- [Background] Katsaros J, Tan E, Zoltie N, Barton M, Venugopalsrinivasan, Venkataramakrishnan. Further experience with the lateral arm free flap. Plast Reconstr Surg. 1991 May;87(5):902-10. doi: 10.1097/00006534-199105000-00015. PMID 2017499
- [Background] Scheker LR, Kleinert HE, Hanel DP. Lateral arm composite tissue transfer to ipsilateral hand defects. J Hand Surg Am. 1987 Sep;12(5 Pt 1):665-72. doi: 10.1016/s0363-5023(87)80045-x. PMID 3309019
- [Background] Wenig BL. The lateral arm free flap for head and neck reconstruction. Otolaryngol Head Neck Surg. 1993 Jul;109(1):116-9. doi: 10.1177/019459989310900121. PMID 8336957
- [Background] Agha RA, Fowler AJ, Rajmohan S, Barai I, Orgill DP; PROCESS Group. Preferred reporting of case series in surgery; the PROCESS guidelines. Int J Surg. 2016 Dec;36(Pt A):319-323. doi: 10.1016/j.ijsu.2016.10.025. Epub 2016 Oct 19. PMID 27770639
- [Background] Sauerbier M, Germann G, Giessler GA, Sedigh Salakdeh M, Doll M. The free lateral arm flap-a reliable option for reconstruction of the forearm and hand. Hand (N Y). 2012 Jun;7(2):163-71. doi: 10.1007/s11552-012-9395-3. PMID 23730235
- [Background] Kuek LB, Chuan TL. The extended lateral arm flap: a new modification. J Reconstr Microsurg. 1991 Jul;7(3):167-73. doi: 10.1055/s-2007-1006775. PMID 1890673
- [Background] Harpf C, Papp C, Ninkovic M, Anderl H, Hussl H. The lateral arm flap: review of 72 cases and technical refinements. J Reconstr Microsurg. 1998 Jan;14(1):39-48. doi: 10.1055/s-2007-1006900. PMID 9524002
- [Background] Klinkenberg M, Fischer S, Kremer T, Hernekamp F, Lehnhardt M, Daigeler A. Comparison of anterolateral thigh, lateral arm, and parascapular free flaps with regard to donor-site morbidity and aesthetic and functional outcomes. Plast Reconstr Surg. 2013 Feb;131(2):293-302. doi: 10.1097/PRS.0b013e31827786bc. PMID 23357991
- [Background] Graham B, Adkins P, Scheker LR. Complications and morbidity of the donor and recipient sites in 123 lateral arm flaps. J Hand Surg Br. 1992 Apr;17(2):189-92. doi: 10.1016/0266-7681(92)90086-h. PMID 1588201
- [Background] Depner C, Erba P, Rieger UM, Iten F, Schaefer DJ, Haug M. Donor-site morbidity of the sensate extended lateral arm flap. J Reconstr Microsurg. 2012 Feb;28(2):133-8. doi: 10.1055/s-0031-1289165. Epub 2011 Sep 29. PMID 21959550